CLINICAL TRIAL: NCT06900790
Title: A Single-Center Retrospective Cohort Study Evaluating the Management and Outcomes of Pediatric Pancreatic Duct Stones Using Endoscopic and Surgical Techniques
Brief Title: Management of Pediatric Pancreatic Calculi At a Single Center: a Retrospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yifan Deng (Other)
Responsible Party: Sponsor-Investigator, Yifan Deng, M.Med, West China Second University Hospital
Organization: West China Second University Hospital (Other)
Other Study IDs: Ethical No. 2024 Review (35)
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Duct Stenting; ERCP; Surgery in Early Childhood; Pediatric Surgery
Keywords: pancreatic duct stones; ERCP; Frey surgery
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ERCP group: Pediatric pancreatic duct stone patients who underwent ERCP to restore pancreatic duct patency.
  Interventions: Procedure: ERCP
- Surgery group: Pediatric pancreatic duct stone patients who underwent Frey surgery.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — There are two intervention methods for pediatric pancreatic duct stones. One is to remove the pancreatic duct stones through Endoscopic Retrograde Cholangiopancreatography(ERCP), while simultaneously dilating the pancreatic duct and placing a stent to assist in the normal drainage of pancreatic juice. The other is local resection of the pancreatic head combined with longitudinal pancreaticojejunostomy (Frey surgery).
  Other Names: Frey surgery

SUMMARY:
The goal of this observational study is to evaluate the long-term effects of ERCP and surgery in pediatric patients with pancreatic duct stones. The main objective is to determine the optimal treatment choice(ERCP or surgery) for children with pancreatic duct stones and identify the appropriate timing for surgery in patients who have undergone multiple ERCP procedures, in order to avoid adverse outcomes caused by repeated trauma to the duodenal papilla.

Last updated on January 24, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 18 years
* Diagnosed with pancreatic duct stones by imaging (e.g., ultrasound, CT, MRCP)
* Treated and followed at pediatric surgery, west china hospital, between 2014 and 2025
* Complete clinical data available for review

Exclusion Criteria:

* Pancreatic duct stones secondary to previous pancreatic or biliary surgery
* Concurrent severe systemic diseases (e.g., advanced cardiac, renal, or hepatic disease)
* Incomplete or missing key clinical records

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents (≤18 years old) diagnosed with pancreatic duct stones between 2015 and 2025 at a single tertiary care center. Data includes patients who underwent ERCP or surgery when the first treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-23 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
stone clearance | From intervention to the end of treatment at 1 week
  The stone clearance rate refers to the proportion of patients confirmed by postoperative imaging (MRCP) to have no residual pancreatic duct stones.
complication rate | From enrollment to the end of treatment at 2 weeks
  The complication rate refers to the incidence of pancreatitis following ERCP and associated procedures, as well as pancreatic fistula, bile leakage, and the necessity for prolonged drainage after the Frey procedure.
reintervention rate | From enrollment to the end of treatment at 1 year.
  The reintervention rate refers to the proportion of patients who required additional invasive procedures (either ERCP or surgery) after the initial treatment.